CLINICAL TRIAL: NCT04467567
Title: Optimization for Clinical Routine of a Dosimetry Protocol Using the Large Field of View VERITON-CT CZT Camera in Patients Treated With LUTATHERA® [177Lu- [DOTA0, Tyr3] -Octreotate
Brief Title: Dosimetry Using a CZT-camera Following LUTATHERA® Therapy
Acronym: EVADOVE177Lu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Elodie CHEVALIER, Principal investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A20200-620
Record Dates: First submitted 2020-06-22; First posted 2020-07-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Dosimetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients treated with lutathera (Experimental): Patients undergoing treatment with Lutathera® and who accept to participate in the study, regardless of the cycle of treatment, 1, 2, 3 or 4.
  Interventions: Other: Single Photon Emission Computed Tomography/ Computed Tomography (SPECT/CT)

INTERVENTIONS:
Other: Single Photon Emission Computed Tomography/ Computed Tomography (SPECT/CT) — SPECT/CT will be performed after Lutathera® treatment (at 24h, 96h and 168h after the infusion of Lutathera®) on the conventional camera and on the VERITON-CT camera

SUMMARY:
The aim of this study is to assess the consistency between a dosimetry protocol using a large field of view CZT-camera and the dosimetry protocol used for recordings acquired with a conventional camera. Therefore, with the conventional camera, recordings are acquired on the "high energy" peak of lutetium 177 (208 keV) using a medium energy collimator. With the VERITON-CT™ CZT camera, recordings are acquired using the low energy peak of 113 keV. A second objective is to compare results between the dosimetry calculated using 3 measurement points (24h, 96h and 168h) and the dosimetry calculated using 2 measurement points (24h and 168h), obtained from the SYMBIA T conventional camera and the VERITON-CT™camera, respectively.

DETAILED DESCRIPTION:
177Lu-DOTATATE has been proven to be an effective therapy for treatment of neuroendocrine tumors. Treatment with [177Lu]-DOTA-TATE consists of 4 cycles, with an infusion of 7.4 GBq (200mCi) every 8 weeks. An imaging protocol to study dosimetry throughout the cycles is essential to determine the average dose absorbed by critical organs and by tumor lesions. The critical organs studied in association with [177Lu]-octreotate treatment are predominantly kidneys and the bone marrow. In this open-label trial, 15 patients undergoing Lutathera® treatment could be enrolled in the study. Patients will have an abdominopelvic SPECT / CT recorded using a conventional Anger camera, followed by a whole-body SPECT / CT recording using a CZT camera. Recordings will be acquired at 24 hours, 96 hours and then at 7 days after the Lutathera® infusion that is administered during one of the 4 treatment cycles. The correlation between the dosimetry results and the appearance of possible grade 3 and 4 side effects will be established.

ELIGIBILITY:
Inclusion Criteria:

* Major adult subject
* ECOG ≤ 2
* Subject receiving treatment with Lutathera®
* Subject having given written, free and informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Contraindication to treatment with Lutathera®
* Subject referred to in articles L. 1121-5, L. 1121-7 and L1121-8 of the public health code.
* Pregnant woman, parturient or nursing mother.
* Subject with a legal protection measure (guardianship, curatorship, safeguard of justice).
* Subject unable to express consent.
* Subject deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care under Articles L. 3212-1 and L.3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Results of the dosimetry obtained from the 2 cameras | 168 hours
  Comparison between dosimetry results obtained from the conventional camera and from the VERITON-CT™ CZT camera.

SECONDARY OUTCOMES:
Results of the dosimetry obtained from the 2 cameras when utilizing 3 points of measurement and when utilizing 2 points of measurement | 24 hours, 96 hours, 168 hours
  Measurement of the average absorbed doses to sensitive organs (bone marrow and kidneys) and to tumor lesions obtained when utilizing 3 measurement points (24h, 96h and 168h) and then obtained when utilizing 2 measurement points (24h and 168h) after the administration of Lutathera®, from both a VERITON-CT™ camera and from a SYMBIA T camera.
Correlation between the dosimetry results | 24 hours, 96 hours, 168 hours
  Average absorbed doses to the kidneys and to the bone marrow versus renal function (creatininaemia, glomerular filtration rate [GFR], blood ionogram), and versus bone marrow activity (blood count).

CONTACTS AND LOCATIONS:
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France